CLINICAL TRIAL: NCT02172495
Title: Tolerability and Efficacy of Spiriva® 18 Micrograms in Patients With COPD in Daily Practice
Brief Title: Spiriva® in Patients With Chronic Obstructive Pulmonary Disease (COPD) in Daily Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.278
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Symptoms of COPD: Patients with symptoms of COPD receiving Tiotropium bromide 18 micrograms
  Interventions: Drug: Tiotropium bromide

INTERVENTIONS:
Drug: Tiotropium bromide — Tiotropium bromide 18 micrograms
  Other Names: Spiriva®

SUMMARY:
Post-marketing surveillance to gather information regarding the tolerance and efficacy of Spiriva® 18 micrograms in patients with COPD under conditions of daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged at least 40 years with the symptoms of Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* Patients with the general and specific contraindications listed in the Patient Information Leaflet and the Basic Product Information

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4700 (Actual)
Dates: Start 2002-06; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in breathlessness when walking/climbing stairs | Baseline, after 4 weeks
Change from baseline in breathlessness on physical exercise | Baseline, after 4 weeks
Change from baseline in breathlessness during everyday activities | Baseline, after 4 weeks
Change from baseline in breathlessness during housework | Baseline, after 4 weeks
Change from baseline in overall severity of the clinical picture | Baseline, after 4 weeks
Occurrence of Adverse Events | 4 weeks